CLINICAL TRIAL: NCT02517944
Title: MYOCARDIAL SILENT INFARCTIONS AND FIBROSIS IN FAMILIAL HYPERCHOLESTEROLEMIA
Brief Title: MYOCARDIAL SILENT INFARCTIONS AND FIBROSIS IN FAMILIAL HYPERCHOLESTEROLEMIA (CHOLCOEUR)
Acronym: CHOLCOEUR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Cardiometabolism and Nutrition, France (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 14DRM_CHOLCOEUR
Record Dates: First submitted 2015-01-14; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Familial Hypercholesterolemia - Heterozygous
Keywords: Familial hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Familial hypercholesterolemia patients: * clinical data
  * biological data
  * cardiac and aortic RMI with gadolinium
- Control group: * clinical data
  * biological data
  * cardiac and aortic RMI with gadolinium

SUMMARY:
Patients with familial hypercholesterolemia (FH) at high cardiovascular risk may suffer from silent micro-infarctions (MI) before clinical coronary heart disease manifestations because of the lifetime exposure to elevated serum LDL-cholesterol levels.

The study aims to demonstrate the higher prevalence of silent myocardial infarction in a population of asymptomatic patients with familial hypercholesterolemia at high cardiovascular risk in comparison to control patients using Cardiac Magnetic Resonance sequences of delayed gadolinium enhancement.

DETAILED DESCRIPTION:
To demonstrate the higher prevalence of silent myocardial infarction in a population of asymptomatic patients with familial hypercholesterolemia at high cardiovascular risk in comparison to control patients, the protocol is the following:

* to enroll 75 patients with familial hypercholesterolemia (FH)
* to enroll 35 subjects without FH (control group)
* for each subject, to collect data from his medical file (blood test results) and to perform a cardiac and aortic MRI in order to evaluate the micro-infarction proportion.

The study will be performed according to GCPs and with respect with french laws.

ELIGIBILITY:
Inclusion criteria:

For patients with heterozygous form of familial hypercholesterolemia:

* Aged between 40 and 60 years
* With an identified genetic mutation (LDL-R, ApoB, PCSK9)
* Asymptomatic,
* With no EKG sign of ischemia
* No personal history of coronary heart disease.
* Treated or untreated by lipid lowering treatment
* High cardiovascular risk identified by 1 of the following criteria:

  1. Current smoking (1 cigarette a day) 2 Family history of very premature onset CHD: first- or second-degree male relative onset before age 45, first- or second-degree female relative onset before age 55 3.Two or more cardiovascular risk factors among this list: increasing age (men > 30, women > 40 years of age), LDL-C > 250 mg/dL, male sex, family history of premature onset CHD, first-degree male relative onset before age 55, first-degree female relative onset before age 65, metabolic syndrome, HDL-C < 40 mg/dL, hypertension (BP > 140/or > 90 mmHg or drug treatment), Lp (a) ≥ 50 mg/dL, tendon xanthoma

For control subjects:

* Aged between 40 and 60 years
* With a normal lipid profile (LDL-C < 1.6g/L HDL-C > 0,45g/L and TG < 4g/L) and untreated by any lipid lowering therapies
* Asymptomatic,
* With EKG showing normal sinus rhythm , no sign of ischemia nor Left Bundle Branch Block
* No personal history of coronary heart disease.
* Control subjects will be matched for age/gender/smoking status and blood pressure

Exclusion criteria:

* Non-affiliation to a healthcare system
* Consent refusal
* Contra-indication to MRI or to gadolinium injection.
* Claustrophobia, metallic devices, pacemaker, mechanical valve implanted before 1985, pregnancy, nursing
* Renal failure
* Technical contra-indication: patient diameter > 70 cm weight > 250 kg
* Personal history of cardiovascular disease and myocardial infarction
* Diabetes mellitus
* Uncontrolled hypertension
* TG < 4 g/L
* Previous use of an Amgen product in the past 12 months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 110 subjects divided into:
  * 75 patients with heterozygous form at high cardiovascular risk
  * 35 controls patients without dyslipidaemia
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients presenting with at least one micro infarction at RMI | Within 4 weeks after consent signature
  Cardiac and aortic RMI with gadolinium

SECONDARY OUTCOMES:
LDL-Cholesterol burden (compared to standard values) | The most recent value within the last 5 years.
Anatomic and functional indexes of the aorta (maximal and minimal areas of aortic lumen, aortic flow) | Within 4 weeks after consent signature
Correlations between LDL-Cholesterol burden & presence of micro infarction, between LDL-Cholesterol burden & myocardial fibrosis, and between LDL-Cholesterol burden & aortic stiffness indexes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenbaum, MD, Principal Investigator — Study principal investigator
Locations (1):
- Unité de prévention des maladies cardiovasculaires- Unité INSERM 939 Pôle Cardiologie/Métabolisme Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Hovingh GK, Davidson MH, Kastelein JJ, O'Connor AM. Diagnosis and treatment of familial hypercholesterolaemia. Eur Heart J. 2013 Apr;34(13):962-71. doi: 10.1093/eurheartj/eht015. Epub 2013 Feb 14. PMID 23416791
- [Background] Nemati MH, Astaneh B. Optimal management of familial hypercholesterolemia: treatment and management strategies. Vasc Health Risk Manag. 2010 Dec 3;6:1079-88. doi: 10.2147/VHRM.S8283. PMID 21191428
- [Background] Descamps OS, Gilbeau JP, Leysen X, Van Leuven F, Heller FR. Impact of genetic defects on atherosclerosis in patients suspected of familial hypercholesterolaemia. Eur J Clin Invest. 2001 Nov;31(11):958-65. doi: 10.1046/j.1365-2362.2001.00915.x. PMID 11737238
- [Background] Austin MA, Hutter CM, Zimmern RL, Humphries SE. Familial hypercholesterolemia and coronary heart disease: a HuGE association review. Am J Epidemiol. 2004 Sep 1;160(5):421-9. doi: 10.1093/aje/kwh237. PMID 15321838
- [Background] Risk of fatal coronary heart disease in familial hypercholesterolaemia. Scientific Steering Committee on behalf of the Simon Broome Register Group. BMJ. 1991 Oct 12;303(6807):893-6. doi: 10.1136/bmj.303.6807.893. PMID 1933004
- [Background] Kroon AA, Ajubi N, van Asten WN, Stalenhoef AF. The prevalence of peripheral vascular disease in familial hypercholesterolaemia. J Intern Med. 1995 Nov;238(5):451-9. doi: 10.1111/j.1365-2796.1995.tb01223.x. PMID 7595185
- [Background] Kolansky DM, Cuchel M, Clark BJ, Paridon S, McCrindle BW, Wiegers SE, Araujo L, Vohra Y, Defesche JC, Wilson JM, Rader DJ. Longitudinal evaluation and assessment of cardiovascular disease in patients with homozygous familial hypercholesterolemia. Am J Cardiol. 2008 Dec 1;102(11):1438-43. doi: 10.1016/j.amjcard.2008.07.035. Epub 2008 Sep 11. PMID 19026292
- [Background] Benn M, Watts GF, Tybjaerg-Hansen A, Nordestgaard BG. Familial hypercholesterolemia in the danish general population: prevalence, coronary artery disease, and cholesterol-lowering medication. J Clin Endocrinol Metab. 2012 Nov;97(11):3956-64. doi: 10.1210/jc.2012-1563. Epub 2012 Aug 14. PMID 22893714
- [Background] Farnier M, Bruckert E. Severe familial hypercholesterolaemia: current and future management. Arch Cardiovasc Dis. 2012 Dec;105(12):656-65. doi: 10.1016/j.acvd.2012.05.011. Epub 2012 Oct 6. PMID 23199621
- [Background] Vilahur G, Casani L, Juan-Babot O, Guerra JM, Badimon L. Infiltrated cardiac lipids impair myofibroblast-induced healing of the myocardial scar post-myocardial infarction. Atherosclerosis. 2012 Oct;224(2):368-76. doi: 10.1016/j.atherosclerosis.2012.07.003. Epub 2012 Jul 22. PMID 22882904
- [Background] Kaufmann PA, Gnecchi-Ruscone T, Schafers KP, Luscher TF, Camici PG. Low density lipoprotein cholesterol and coronary microvascular dysfunction in hypercholesterolemia. J Am Coll Cardiol. 2000 Jul;36(1):103-9. doi: 10.1016/s0735-1097(00)00697-5. PMID 10898420
- [Background] Dayanikli F, Grambow D, Muzik O, Mosca L, Rubenfire M, Schwaiger M. Early detection of abnormal coronary flow reserve in asymptomatic men at high risk for coronary artery disease using positron emission tomography. Circulation. 1994 Aug;90(2):808-17. doi: 10.1161/01.cir.90.2.808. PMID 8044952
- [Background] Giulia Gagliardi M, Crea F, Polletta B, Bassano C, La Vigna G, Ballerini L, Ragonese P. Coronary microvascular endothelial dysfunction in transplanted children. Eur Heart J. 2001 Feb;22(3):254-60. doi: 10.1053/euhj.2001.2105. PMID 11161937
- [Background] Watts GF, Sullivan DR, Poplawski N, van Bockxmeer F, Hamilton-Craig I, Clifton PM, O'Brien R, Bishop W, George P, Barter PJ, Bates T, Burnett JR, Coakley J, Davidson P, Emery J, Martin A, Farid W, Freeman L, Geelhoed E, Juniper A, Kidd A, Kostner K, Krass I, Livingston M, Maxwell S, O'Leary P, Owaimrin A, Redgrave TG, Reid N, Southwell L, Suthers G, Tonkin A, Towler S, Trent R; Familial Hypercholesterolaemia Australasia Network Consensus Group (Australian Atherosclerosis Society). Familial hypercholesterolaemia: a model of care for Australasia. Atheroscler Suppl. 2011 Oct;12(2):221-63. doi: 10.1016/j.atherosclerosissup.2011.06.001. Epub 2011 Sep 13. PMID 21917530
- [Background] De Backer G, Ambrosioni E, Borch-Johnsen K, Brotons C, Cifkova R, Dallongeville J, Ebrahim S, Faergeman O, Graham I, Mancia G, Cats VM, Orth-Gomer K, Perk J, Pyorala K, Rodicio JL, Sans S, Sansoy V, Sechtem U, Silber S, Thomsen T, Wood D; European Society of Cardiology. American Heart Association. American College of Cardiology. European guidelines on cardiovascular disease prevention in clinical practice. Third Joint Task Force of European and other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of eight societies and by invited experts). Atherosclerosis. 2004 Apr;173(2):381-91. No abstract available. PMID 15195638
- [Background] Nordestgaard BG, Chapman MJ, Humphries SE, Ginsberg HN, Masana L, Descamps OS, Wiklund O, Hegele RA, Raal FJ, Defesche JC, Wiegman A, Santos RD, Watts GF, Parhofer KG, Hovingh GK, Kovanen PT, Boileau C, Averna M, Boren J, Bruckert E, Catapano AL, Kuivenhoven JA, Pajukanta P, Ray K, Stalenhoef AF, Stroes E, Taskinen MR, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Familial hypercholesterolaemia is underdiagnosed and undertreated in the general population: guidance for clinicians to prevent coronary heart disease: consensus statement of the European Atherosclerosis Society. Eur Heart J. 2013 Dec;34(45):3478-90a. doi: 10.1093/eurheartj/eht273. Epub 2013 Aug 15. PMID 23956253
- [Background] Kwong RY, Sattar H, Wu H, Vorobiof G, Gandla V, Steel K, Siu S, Brown KA. Incidence and prognostic implication of unrecognized myocardial scar characterized by cardiac magnetic resonance in diabetic patients without clinical evidence of myocardial infarction. Circulation. 2008 Sep 2;118(10):1011-20. doi: 10.1161/CIRCULATIONAHA.107.727826. Epub 2008 Aug 25. PMID 18725488
- [Background] Mewton N, Liu CY, Croisille P, Bluemke D, Lima JA. Assessment of myocardial fibrosis with cardiovascular magnetic resonance. J Am Coll Cardiol. 2011 Feb 22;57(8):891-903. doi: 10.1016/j.jacc.2010.11.013. PMID 21329834
- [Background] Choi DS, Ha JW, Choi B, Yang WI, Choi EY, Rim SJ, Chung N. Extent of late gadolinium enhancement in cardiovascular magnetic resonance and its relation with left ventricular diastolic function in patients with hypertrophic cardiomyopathy. Circ J. 2008 Sep;72(9):1449-53. doi: 10.1253/circj.cj-07-0874. PMID 18724020
- [Background] Lin Y, Yang SG, Chen H, Zhang HQ, Wang CS. [The predictive value of DE-CMR in patients with severe chronic aortic regurgitation and extremely dilated left ventricular chamber]. Zhonghua Wai Ke Za Zhi. 2012 Dec;50(12):1087-90. Chinese. PMID 23336485
- [Background] Kuruvilla S, Adenaw N, Katwal AB, Lipinski MJ, Kramer CM, Salerno M. Late gadolinium enhancement on cardiac magnetic resonance predicts adverse cardiovascular outcomes in nonischemic cardiomyopathy: a systematic review and meta-analysis. Circ Cardiovasc Imaging. 2014 Mar;7(2):250-258. doi: 10.1161/CIRCIMAGING.113.001144. Epub 2013 Dec 20. PMID 24363358
- [Background] Lipinski MJ, McVey CM, Berger JS, Kramer CM, Salerno M. Prognostic value of stress cardiac magnetic resonance imaging in patients with known or suspected coronary artery disease: a systematic review and meta-analysis. J Am Coll Cardiol. 2013 Aug 27;62(9):826-38. doi: 10.1016/j.jacc.2013.03.080. Epub 2013 May 30. PMID 23727209
- [Background] Mascherbauer J, Marzluf BA, Tufaro C, Pfaffenberger S, Graf A, Wexberg P, Panzenbock A, Jakowitsch J, Bangert C, Laimer D, Schreiber C, Karakus G, Hulsmann M, Pacher R, Lang IM, Maurer G, Bonderman D. Cardiac magnetic resonance postcontrast T1 time is associated with outcome in patients with heart failure and preserved ejection fraction. Circ Cardiovasc Imaging. 2013 Nov;6(6):1056-65. doi: 10.1161/CIRCIMAGING.113.000633. Epub 2013 Sep 13. PMID 24036385
- [Background] Dall'Armellina E, Ferreira VM, Kharbanda RK, Prendergast B, Piechnik SK, Robson MD, Jones M, Francis JM, Choudhury RP, Neubauer S. Diagnostic value of pre-contrast T1 mapping in acute and chronic myocardial infarction. JACC Cardiovasc Imaging. 2013 Jun;6(6):739-42. doi: 10.1016/j.jcmg.2012.11.020. No abstract available. PMID 23764100
- [Background] Liu CY, Liu YC, Wu C, Armstrong A, Volpe GJ, van der Geest RJ, Liu Y, Hundley WG, Gomes AS, Liu S, Nacif M, Bluemke DA, Lima JAC. Evaluation of age-related interstitial myocardial fibrosis with cardiac magnetic resonance contrast-enhanced T1 mapping: MESA (Multi-Ethnic Study of Atherosclerosis). J Am Coll Cardiol. 2013 Oct 1;62(14):1280-1287. doi: 10.1016/j.jacc.2013.05.078. Epub 2013 Jul 17. PMID 23871886
- [Background] Sacre K, Brihaye B, Hyafil F, Serfaty JM, Escoubet B, Zennaro MC, Lidove O, Laissy JP, Papo T. Asymptomatic myocardial ischemic disease in antiphospholipid syndrome: a controlled cardiac magnetic resonance imaging study. Arthritis Rheum. 2010 Jul;62(7):2093-100. doi: 10.1002/art.27488. PMID 20506512
- [Background] Cheng HM, Ye ZX, Chiou KR, Lin SJ, Charng MJ. Vascular stiffness in familial hypercholesterolaemia is associated with C-reactive protein and cholesterol burden. Eur J Clin Invest. 2007 Mar;37(3):197-206. doi: 10.1111/j.1365-2362.2007.01772.x. PMID 17359487
- [Background] Schmidt HH, Hill S, Makariou EV, Feuerstein IM, Dugi KA, Hoeg JM. Relation of cholesterol-year score to severity of calcific atherosclerosis and tissue deposition in homozygous familial hypercholesterolemia. Am J Cardiol. 1996 Mar 15;77(8):575-80. doi: 10.1016/s0002-9149(97)89309-5. PMID 8610605